CLINICAL TRIAL: NCT04015245
Title: Benefits of SNMC (Stronger Neo-Minophagen C ) for Heptoma Patient With Acute Hepatitis Post Transarterial Chemoembolization Therapy
Brief Title: SNMC (Stronger Neo-Minophagen C ) for Acute Hepatitis Post Transarterial Chemoembolization Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chimei Medical Center (Other)
Responsible Party: Principal Investigator, Hsing-Tao Kuo, attending physician, Chimei Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CMMC10702-001
Record Dates: First submitted 2019-05-28; First posted 2019-07-10 (Actual); Last update posted 2019-07-10 (Actual); Status verified 2019-07

CONDITIONS: Hepatocellular Carcinoma
Keywords: TACE
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — stronger neominophagen C

STUDY DESIGN:
Intervention Model Description: randomized control trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SNMC (Experimental)
  Interventions: Drug: Stronger Neo-Minophagen C
- non-SNMC (No Intervention)

INTERVENTIONS:
Drug: Stronger Neo-Minophagen C — intravenous injection after TACE
  Arms: SNMC

SUMMARY:
A glycyrrhizin-containing product, Stronger Neo-Minophagen C TM (SNMC; Minophagen Pharmaceutical Co.Ltd.,Tokyo,Japan),is widely used in Japan for suppression of hepatitis activity and for prevention of disease progression in patients with hepatitis B virus- and HCV-induced chronic hepatitis. In Taiwan, SNMC has been licensed by Taiwan Food and Drug Administration for the indication of maintain hepatic function. Glycyrrhizin has been reported to mitigate hepatic inflammation by suppressing elevated alanine aminotransferase(ALT) levels and preventing disease progression. The effect of SNMC on acute deterioration of hepatic function following transarterial chemoembolization (TACE) was still unknown. This study aimed to evaluate the effect of SNMC on acute deterioration of hepatic function following TACE.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is the fifth most common cancer in the world and the most common primary liver cancer. There are a variety of therapies for treatment of HCC; among them, transarterial chemoembolization (TACE) is one of the most commonly used treatment modalities. TACE induces ischemic tumor necrosis by obstruction of hepatic artery blood flow and exerts an anticancer effect via chemotherapeutic agents such as adriamycin or cisplatin mixed with Lipiodol. In the American Association for the Study of Liver Diseases (AASLD) guidelines for the management of HCC, TACE is recommended for patients with intermediate-stage HCC according to the Barcelona Clinic Liver Cancer (BCLC) staging system, because TACE was found to improve survival compared with the best supportive care in patients with unresectable HCC. Although TACE is the established standard of care only for intermediate-stage HCC, in recent years, TACE has been used widely even in treatment of advanced-stage HCC. The most frequent side effects of TACE are fever, nausea, and abdominal pain, and these side effects are self-limiting in the majority of patients. However, acute deterioration of hepatic function following TACE is a potentially life-threatening complication that occasionally interferes with continuation of TACE in patients with HCC. Although TACE has marked direct antitumor effects, it can also result in more complications than conservative management, because the ischemic damage caused by TACE can influence not only tumor tissue but non-tumorous liver tissue.This study aimed to evaluate the effect of SNMC on acute deterioration of hepatic function following TACE.

ELIGIBILITY:
Inclusion Criteria:

1. Intermediate-stage HCC according to the Barcelona Clinic Liver Cancer (BCLC) staging system, either treatment naïve or experienced.
2. Child's score belong to A or B(7)
3. Total bilirubin level <2 and Prothrombin time prolong <3"

Exclusion Criteria:

1. Had history of liver decompensation (ascites, encephalopathy, jaundice and varices bleeding) before this TACE
2. has allergic history of SNMC
3. consensus form cannot be available
4. hypokalemia (<3.5 mmol/L)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-04-12 (Actual); Primary Completion 2019-05-09 (Actual); Study Completion 2019-05-28 (Actual)

PRIMARY OUTCOMES:
Series changes of serum levels of alanine aminotransferase | 4 days
  To evaluate the daily change of serum levels of alanine aminotransferase before and after TACE, which indicate the hepatitis activity caused by TACE
Series changes of serum levels of aspartate aminotransferase | 4 days
  To evaluate the daily change of serum levels of aspartate aminotransferase before and after TACE, which indicate the hepatitis activity caused by TACE
Series changes of serum levels of Total bilirubin | 4 days
  To evaluate the daily change of serum levels of Total bilirubin before and after TACE, which indicate the hepatitis activity caused by TACE
Series changes of Prothrombin Time | 4 days
  To evaluate the daily change of Prothrombin Time before and after TACE, which indicate the hepatitis activity caused by TACE
Series changes of Prothrombin Time-Intemrnational Normalized Ratio | 4 days
  To evaluate the daily change of Series changes of Prothrombin Time-Intemrnational Normalized Ratio before and after TACE, which indicate the hepatitis activity caused by TACE

SECONDARY OUTCOMES:
Series changes of potassium levels before and after TACE | 4 days
  To evaluate the daily change of Series changes of potassium levels before and after TACE, which indicate the side effect caused by SNMC
Series changes of blood pressure levels before and after TACE | 4 days
  To evaluate the daily change of Series changes of blood pressure levels before and after TACE, which indicate the side effect caused by SNMC

CONTACTS AND LOCATIONS:
Locations (1):
- ChiMei Medical Center, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No